CLINICAL TRIAL: NCT03419988
Title: Cell Signaling and Resistance to Oxidative Stress: Effects of Aging and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Arizona University (Other)
Responsible Party: Principal Investigator, Tinna Traustadottir, Associate Professor, Biological Sciences, Northern Arizona University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R15AG055077 (NIH)
Record Dates: First submitted 2018-01-11; First posted 2018-02-05 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Aging
Keywords: Nrf2

STUDY DESIGN:
Intervention Model Description: Randomized control trial: exercise intervention versus non-exercise control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): 8-weeks exercise intervention: 3-days per week for 45-55 minutes per session
  Interventions: Behavioral: Exercise Intervention
- Control (No Intervention): 8-weeks control: asked not to change anything or start exercising.

INTERVENTIONS:
Behavioral: Exercise Intervention — 24 sessions of aerobic exercise
  Arms: Exercise Intervention

SUMMARY:
Advanced age is the main risk factor for chronic diseases such as cardiovascular disease, type 2 diabetes, Alzheimer's disease and cancer. One reason may be due to decreased resistance to oxidative stress as antioxidant defenses and cell protection is reduced with aging. This has been shown in animal studies and also that the impairment can be somewhat restored with exercise. This will be the first study to test this in humans by comparing young and older inactive adults before and after an exercise intervention, a practical and cost-effective intervention that can have tremendous public health impact by lowering risk for disease and medical-related costs.

DETAILED DESCRIPTION:
Advanced age substantially increases the risk for a host of diseases including cardiovascular disease, type 2 diabetes, Alzheimer's disease, and cancer. A major factor that appears to underlie this increased risk with age is reduced capacity to resist oxidative injury or oxidative stress. Therefore, maintaining or increasing the capacity to resist oxidative stress appears critical to the prevention of age-related disease and promotion of successful aging. One potential reason for the lower resistance to oxidative stress with age is a gradual shift in the redox state toward a more oxidized cellular environment potentially disrupting cell-signaling. Nuclear erythroid-2-p45-related factor-2 (Nrf2) is the master regulator of antioxidant defenses. Nrf2 drives expression of a host of genes involved in cellular detoxification and antioxidant defenses. There is strong evidence from animal studies that Nrf2 signaling is reduced with aging and can be at least partially restored with moderate exercise training, however the gap in current knowledge is whether these data do in fact translate to humans. This study will test the following hypotheses in young and older men and women: i) aging is associated with impaired Nrf2 signaling in response to acute exercise and ii) moderate exercise training will improve Nrf2 signaling in older, inactive individuals, and this will increase their resistance to oxidative stress. These hypotheses will be tested by comparing 25 young (18-28y) and 25 older (≥60y) inactive individuals before and after an 8-week exercise intervention (n=15 per age group) and in comparison to non-exercising age-matched control groups (n=10 per age group). Nrf2 signaling will be measured in peripheral blood mononuclear cells (PBMCs) in response to acute exercise and will include gene expression (NRF2, NQO1, HO1, GCLC), protein abundance (NRF2, KEAP1, NQO1, HO1, GCLC) and Nrf2-ARE binding capacity. Resistance to oxidative stress will be measured by plasma F2-isoprostane response to forearm ischemia/reperfusion. The results will increase understanding of the mechanisms of diminished stress resilience with aging and the plasticity of these pathways. This will determine whether targeting Nrf2 signaling will be effective for prevention or treatment of these age-related changes which has an enormous public health impact due to the potential of lowering disease risk and medical costs. An additional significance of this project is creating opportunity for undergraduate and graduate students to become involved in research, an important purpose of the Academic Research Enhancement Award (AREA) program and a mission of Northern Arizona University.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-28 years or 60 years and older
* Competent to independently give informed consent
* Successful completion of screening
* No regular exercise for the past 6-months (by self-report)
* A score below 3.0 on the Historical Lifetime Physical Activity Questionnaire

Exclusion Criteria:

* Estrogen supplementation within the previous 6 months
* Use of anti-oxidant supplements, in excess of standard multi-vitamins (1 tablet/day)
* Current smoker
* Body Mass Index (BMI) ≤33 kg/m2 (Class I Obesity)
* Any chronic illness that could affect outcome measures, including diabetes, liver or renal disease, or cancer (other than skin cancer)
* History of a myocardial infarction within the last 6 months, clinically significant aortic stenosis, use of cardiac defibrillator, or uncontrolled angina
* Clinically significant arrhythmia on a resting EKG or significant EKG changes during the baseline maximal oxygen consumption (VO2 max) test
* Any other condition that would contraindicate maximal exercise testing, including elevated blood pressure at rest (systolic BP >150 or diastolic BP >90 mm Hg on at least 2 measurements, at least 10 minutes apart) or musculoskeletal problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Cell signaling | 8 weeks
  Nuclear Nrf2 protein content in peripheral mononuclear cells (PBMCs) in response to acute exercise
Resistance to oxidative stress | 8 weeks
  F2-isoprostane response to forearm ischemia-reperfusion

SECONDARY OUTCOMES:
Cell signaling | 8 weeks
  GCLC protein abundance in PBMCs in response to acute exercise

CONTACTS AND LOCATIONS:
Overall Officials: Tinna Traustadóttir, PhD, Principal Investigator — Northern Arizona University
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ostrom EL, Traustadottir T. Aerobic exercise training partially reverses the impairment of Nrf2 activation in older humans. Free Radic Biol Med. 2020 Nov 20;160:418-432. doi: 10.1016/j.freeradbiomed.2020.08.016. Epub 2020 Aug 28. PMID 32866619